CLINICAL TRIAL: NCT01378975
Title: An Open-label, Single-arm, Phase II, Multicenter Study, to Evaluate the Efficacy of Vemurafenib in Metastatic Melanoma Patients With Brain Metastases
Brief Title: A Study of Vemurafenib in Metastatic Melanoma Participants With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO25743
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

ARMS (2):
- Cohort 1: Previously Untreated Participants (Experimental): Participants who had not received previous treatment for brain metastases [i.e., had never received brain stereotactic radiotherapy (SRT), whole-brain radiotherapy (WBRT), surgery, or any other treatment for their brain metastases] received Vemurafenib 960 milligram (mg) tablet orally, twice daily (BID) from Day 1 until development of progressive disease within the brain or outside of the brain (whichever occurred first), unacceptable toxicity, consent withdrawal, protocol violation endangering participant's safety, death, reasons deemed by the investigator, or study termination by the Sponsor.
  Interventions: Drug: Vemurafenib
- Cohort 2: Previously treated Participants (Experimental): Participants who were previously treated with brain SRT, WBRT, or surgery for their brain metastases and have progressed following this treatment, received Vemurafenib 960 milligram (mg) tablet orally, BID from Day 1 until development of progressive disease within the brain or outside of the brain (whichever occurred first), unacceptable toxicity, consent withdrawal, protocol violation endangering participant's safety, death, reasons deemed by the investigator, or study termination by the Sponsor.
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — 960 mg oral doses twice daily until disease progression, unacceptable toxicity or consent withdrawal.

SUMMARY:
This open-label, single-arm, multicenter study will evaluate the efficacy and safety in participants with metastatic melanoma who developed brain metastases. Participants may or may not have received prior systemic treatment for metastatic melanoma [except treatment with v-raf murine sarcoma viral oncogene homolog B (BRAF) or mitogen-activated protein kinase (MEK) inhibitors]. Participants will receive oral doses of 960 mg vemurafenib twice daily until disease progression, unacceptable toxicity or consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Histologically confirmed metastatic melanoma (Stage IV, American Joint Committee on Cancer) with BRAF V600 mutation (cobas 4800 BRAF V600 Mutation Test)
* Measurable brain metastases, defined as lesions that were accurately measured in at least one dimension (longest diameter to be recorded) as ≥0.5 cm in the brain MRI with contrast, treated or untreated
* Participants may or may not have received prior systemic therapy for metastatic melanoma and either a) have received no prior treatment for brain metastases or b) have received prior treatment for brain metastases and have progressed
* Participants may or may not have symptoms related to their brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Participants must have recovered from all side effects of their most recent systemic or local treatment for metastatic melanoma

Exclusion Criteria:

* Increasing corticosteroid dose during the 7 days prior to first dose of study drug
* Leptomeningeal involvement in participants with no prior treatment for brain metastases
* Previous malignancy requiring active treatment within the past 2 years, except for treated and controlled basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix
* Concurrent administration of any anticancer therapies other than those administered in the study
* Treatment with any cytotoxic, investigational drug or targeted therapy 4 weeks prior to first dose of study drug. Radiation therapy ≤1 week prior to first administration of vemurafenib; and stereotactic radiotherapy ≤1 day prior to prior to first administration of vemurafenib
* Prior treatment with BRAF or MEK inhibitors
* Clinically significant cardiovascular disease or event within the 6 months prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (10):
  - Los Angeles, California
  - Aurora, Colorado
  - Tampa, Florida
  - Boston, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Charlotte, North Carolina
  - Dallas, Texas
  - Seattle, Washington
- Australia (2):
  - Wentworthville, New South Wales
  - Melbourne, Victoria
- Toronto, Ontario, Canada
- France (3):
  - Bordeaux
  - Nice
  - Paris
- Germany (6):
  - Essen
  - Frankfurt
  - Kiel
  - Mannheim
  - Münster
  - Tübingen
- Tel Litwinsky, Israel
- Italy (2):
  - Milan, Lombardy
  - Siena, Tuscany
- Netherlands (2):
  - Amsterdam
  - Groningen
- Spain (3):
  - Pamplona, Navarre
  - Barcelona
  - Madrid
- Northwood, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Started | 90 | 56
Completed | 4 | 6
Not Completed | 86 | 50
Not completed — Death | 77 | 46
Not completed — Investigator Request | 1 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrew Consent | 4 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants | Total
Number analyzed (Participants) | 90 | 56 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (12.73) | 52.7 (13.85) | 54.5 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 22 | 56
  Male | 56 | 34 | 90

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (BORR) Within Brain of Previously Untreated Participants (Assessed by Independent Review Committee [IRC] Using Modified Response Evaluation Criteria in Solid Tumors [RECIST])
Description: BORR assessed by IRC is defined as percentage of participants who were responders [with best overall response (BOR) documented as confirmed complete response (CR) or partial response (PR)]. The RECIST v1.1 criteria modified for independent review of body and brain lesions was based on current radiology practices. The modifications to RECIST v1.1 included allowing target lesions in the brain to be >=5 mm by contrast-enhanced magnetic resonance imaging scan (in traditional RECIST v1.1 this is >=10 mm), allowing up to 5 target lesions in the brain (in traditional RECIST v1.1 only 2 target lesions), and examining the lesions within the brain and outside the brain separately for analytical purposes. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm), PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The intent to treat (ITT) population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Previously Untreated Participants
Number analyzed (Participants) | 90
percentage of participants | 17.8 [10.5 to 27.3]

2. Secondary Outcome: Best Overall Response Rate (BORR) in the Brain of Participants With Previously Treated or Untreated Brain Metastases as Assessed by the IRC Using RECIST v1.1
Description: Percentage of participants who were responders with BOR documented as confirmed CR or PR, stable disease (SD), progressive disease (PD). CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 90 | 56
percentage of participants
  Complete Response | 2.2 | 0.0
  Partial Response | 15.6 | 17.9
  Stable Disease | 43.3 | 41.1
  Progressive Disease | 32.2 | 33.9
  Unevaluable | 6.7 | 7.1

3. Secondary Outcome: Best Overall Response Rate (BORR) in the Brain of Participants With Previously Treated Brain Metastases as Assessed by the IRC Using RECIST v1.1
Description: BORR within brain assessed by IRC is defined as percentage of participants who were responders (with BOR documented as confirmed CR or PR). According to RECIST v1.1 criteria modified for brain metastases, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 56
percentage of participants | 17.9 [8.9 to 30.4]

4. Secondary Outcome: Best Overall Response Rate Outside the Brain (Assessed by IRC)
Description: BORR outside of brain assessed by IRC is defined as percentage of participants who were responders (with BOR documented as confirmed CR or PR). According to RECIST v1.1 criteria modified for brain metastases, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm, PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study. Here, number participants analyzed is the total number of participants who had measurable disease outside brain at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 79 | 40
percentage of participants | 32.9 [22.7 to 44.4] | 22.5 [10.8 to 38.5]

5. Secondary Outcome: Duration of Response (DOR) (Assessed by Investigator and IRC)
Description: Duration of response was defined as the time interval between the date of the earliest qualifying response and the earliest date of PD or death from any cause. For participants who were alive without progression following the qualifying response, DOR were censored on the date of last available tumor assessment on or before the data cutoff date.
Time Frame: Date of the earliest qualifying response until the earliest date of PD or death from any cause (approximately up to 4 years)
Population: The ITT population included all participants who were enrolled in the study. Here, 'n' indicates number of participants who were responders within brain or outside brain assessed by investigator or IRC.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 26 | 13
months
  Investigator: DOR (Within Brain) (n=26, 13) | 4.67 [2.66 to 24.21] | 6.64 [1.87 to 21.98]
  Investigator: DOR (Outside Brain) (n=25, 11): number analyzed (Participants) | 25 | 11
  Investigator: DOR (Outside Brain) (n=25, 11) | 5.55 [1.84 to 25.63] | 10.74 [1.84 to 23.10]
  IRC: DOR (Within Brain) (n=16, 10): number analyzed (Participants) | 16 | 10
  IRC: DOR (Within Brain) (n=16, 10) | 4.60 [2.66 to 29.90] | 6.64 [0.95 to 18.40]
  IRC: DOR (Outside Brain) (n=26, 9): number analyzed (Participants) | 26 | 9
  IRC: DOR (Outside Brain) (n=26, 9) | 7.72 [1.84 to 21.55] | 11.07 [1.84 to 23.10]

6. Secondary Outcome: Progression-Free Survival (PFS) Based on Overall Tumor Response (Assessed by Investigator)
Description: Progression-free survival was defined as the time between enrollment on Day 1 and the date of first radiographically documented progressive disease (within or outside the brain), clinical progressive disease, as assessed by the investigator or death whichever occurred first.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 90 | 56
months | 3.65 [0.30 to 33.35] | 3.71 [0.26 to 27.37]

7. Secondary Outcome: Progression-Free Survival (PFS) Based on Tumor Assessment Within Brain Only (Assessed by Investigator )
Description: Progression-free survival was defined as the time between enrollment on Day 1 and the date of first radiographically documented progressive disease (within brain), clinical progressive disease, as assessed by the investigator or death whichever occurred first.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 90 | 56
months | 3.68 [0.36 to 33.35] | 4.04 [0.26 to 27.37]

8. Secondary Outcome: Time to Development of New Brain Metastases in Responders
Description: Time to development of new lesions within the brain was defined as the interval between the date of first treatment and the earliest date of documentation of new brain lesions. Participants who were known to be free of new lesions were censored on the date of last tumor assessment.
Time Frame: Date of first treatment and the earliest date of documentation of new brain lesions (approximately up to 4 years)
Population: The ITT population included all participants who were enrolled in the study. Here, number of participants analyzed is the participants who were responders.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 26 | 13
months | 14.92 [3.48 to 33.35] | 14.52 [2.79 to 27.37]

9. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time between enrollment on Day 1 and date of death, irrespective of the cause of death. Participants for whom no death was captured on the clinical database were censored at the latest date they were known to be alive prior to or on the cutoff date.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 90 | 56
months | 8.87 [0.59 to 34.53] | 9.63 [0.66 to 34.30]

10. Secondary Outcome: Best Overall Response Rate (BORR) Within the Brain and Outside Brain (Assessed by Investigator)
Description: as for outcome 2
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study. Here, 'n' indicates the number participants who were evaluable for within brain assessment and who had measurable disease outside brain at baseline for outside brain assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 90 | 56
percentage of participants
  Complete Response (Within Brain) (n=90, 56) | 2.2 | 0.0
  Partial Response (Within Brain) (n=90, 56) | 26.7 | 23.2
  Stable Disease (Within Brain) (n=90, 56) | 40.0 | 53.6
  Progressive Disease (Within Brain) (n=90, 56) | 27.8 | 19.6
  Unevaluable (Within Brain) (n=90, 56) | 3.3 | 3.6
  Complete Response (Outside Brain) (n=79, 40): number analyzed (Participants) | 79 | 40
  Complete Response (Outside Brain) (n=79, 40) | 0.0 | 5.0
  Partial Response (Outside Brain) (n=79, 40): number analyzed (Participants) | 79 | 40
  Partial Response (Outside Brain) (n=79, 40) | 31.6 | 22.5
  Stable Disease (Outside Brain) (n=79, 40): number analyzed (Participants) | 79 | 40
  Stable Disease (Outside Brain) (n=79, 40) | 49.4 | 52.5
  Progressive Disease (Outside Brain) (n=79, 40): number analyzed (Participants) | 79 | 40
  Progressive Disease (Outside Brain) (n=79, 40) | 11.4 | 15.0
  Unevaluable (Outside Brain) (n=79, 40): number analyzed (Participants) | 79 | 40
  Unevaluable (Outside Brain) (n=79, 40) | 7.6 | 5.0

11. Secondary Outcome: Best Overall Response Rate (BORR) Within the Brain and Outside Brain (Not Necessarily Follows the RECIST Criteria - as Assessed by Investigator)
Description: Percentage of participants who were responders (with best overall response (BOR) documented as confirmed complete response [CR] or partial response [PR]) were reported.
Time Frame: Baseline up to the disease progression or death from any cause (approximately 4 years)
Population: The ITT population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 90 | 56
percentage of participants | 18.9 [11.4 to 28.5] | 17.9 [8.9 to 30.4]

12. Secondary Outcome: Percentage of Participants With Adverse Events (AE)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: From signing of informed consent form up to 28 days after the last dose of study drug (approximately up to 4 years)
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
Number analyzed (Participants) | 90 | 56
percentage of participants | 97.8 | 94.6

ADVERSE EVENTS:
Time Frame: From signing of informed consent form up to 28 days after the last dose of study drug (Up to approximately 4 years)
Description: The safety population included all participants who received at least one dose of study medication.
Arm/Group | Cohort 1: Previously Untreated Participants | Cohort 2: Previously Treated Participants
All-Cause Mortality (participants affected / at risk) | 77/90 | 46/56
Serious Adverse Events (participants affected / at risk) | 37/90 | 27/56
Other Adverse Events (participants affected / at risk) | 85/90 | 53/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Previously Untreated Participants (N=90) | Cohort 2: Previously Treated Participants (N=56)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 6
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsillar neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Abscess rupture (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 1
Ocular ischaemic syndrome (Eye disorders) | 0 | 1
Papilloedema (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Previously Untreated Participants (N=90) | Cohort 2: Previously Treated Participants (N=56)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 28 | 13
Rash (Skin and subcutaneous tissue disorders) | 29 | 17
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 18 | 17
Erythema (Skin and subcutaneous tissue disorders) | 13 | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 10
Actinic keratosis (Skin and subcutaneous tissue disorders) | 6 | 5
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 9 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 4 | 3
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 3
Fatigue (General disorders) | 22 | 19
Asthenia (General disorders) | 13 | 6
Oedema peripheral (General disorders) | 7 | 8
Pyrexia (General disorders) | 11 | 7
Pain (General disorders) | 6 | 5
Chest Pain (General disorders) | 1 | 4
Xerosis (General disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Electrocardiogram QT prolonged (Investigations) | 22 | 8
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood bilirubin increased (Investigations) | 6 | 4
Alanine aminotransferase increased (Investigations) | 6 | 5
Blood alkaline phosphatase increased (Investigations) | 5 | 2
Weight decreased (Investigations) | 6 | 6
Blood creatinine increased (Investigations) | 5 | 3
Nausea (Gastrointestinal disorders) | 15 | 14
Diarrhoea (Gastrointestinal disorders) | 14 | 10
Vomoting (Gastrointestinal disorders) | 8 | 8
Constipation (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Faecal incontinence (Gastrointestinal disorders) | 0 | 3
Headache (Nervous system disorders) | 16 | 8
Paraesthesia (Nervous system disorders) | 9 | 2
Dysgeusia (Nervous system disorders) | 6 | 4
Seizure (Nervous system disorders) | 2 | 6
Dizziness (Nervous system disorders) | 3 | 3
Balance disorder (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 0 | 5
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 12
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Nasopharyngitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 4
Conjunctivitis (Infections and infestations) | 2 | 3
Folliculitis (Infections and infestations) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 5 | 7
Confusional state (Psychiatric disorders) | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 8 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5
Hypertension (Vascular disorders) | 6 | 4
Photophobia (Eye disorders) | 2 | 3
Visual impairment (Eye disorders) | 1 | 3
Sunburn (Injury, poisoning and procedural complications) | 6 | 2
Contrast media allergy (Immune system disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.